CLINICAL TRIAL: NCT00000251
Title: Effects of Subanesthetic Concentrations of Isoflurane/Nitrous Oxide
Brief Title: Effects of Subanesthetic Concentrations of Isoflurane/Nitrous Oxide - 3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NIDA-08391-3; R01DA008391 (NIH); R01-08391-3
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: nitrous oxide; isoflurane; subjective effects; psychomotor; healthy volunteer; drug interaction
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Isoflurane; Oxygen

STUDY DESIGN:
Who Masked: Participant

ARMS (6):
- Placebo (Placebo Comparator): Subjects inhale 100% oxygen
  Interventions: Other: 100% oxygen
- 30% N2O (Active Comparator): Subjects inhale 30% N2O
  Interventions: Drug: 30% N2O
- 0.2% isoflurane (Active Comparator): Subjects inhale 0.2% isoflurane
  Interventions: Drug: 0.2% isoflurane
- 0.4% isoflurane (Active Comparator): Subjects inhale 0.4% isoflurane
  Interventions: Drug: 0.4% isoflurane
- 0.2% isoflurane + 30% N2O (Active Comparator): Subjects will inhale a combination of 0.2% isoflurane and 30% N2O
  Interventions: Drug: 30% N2O; Drug: 0.2% isoflurane
- 0.4% isoflurane + 30% N2O (Active Comparator): Subjects will inhale a combination of 0.4% isoflurane and 30% N2O
  Interventions: Drug: 30% N2O; Drug: 0.4% isoflurane

INTERVENTIONS:
Drug: 30% N2O
  Arms: 0.2% isoflurane + 30% N2O; 0.4% isoflurane + 30% N2O; 30% N2O
Drug: 0.2% isoflurane
  Arms: 0.2% isoflurane; 0.2% isoflurane + 30% N2O
Drug: 0.4% isoflurane
  Arms: 0.4% isoflurane; 0.4% isoflurane + 30% N2O
Other: 100% oxygen — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to conduct experiments to examine subjective and reinforcing effects of nitrous oxide. Mood altering and psychomotor effects will be tested on non-drug abusers and preference procedures will be used to assess reinforcing effects. To evaluate the acute and residual effects of subanesthetic concentrations of isoflurane/nitrous oxide combinations in healthy volunteers.

ELIGIBILITY:
Please contact site for information.

Ages: 21 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 1994-04; Primary Completion 1996-01 (Actual); Study Completion 1996-01 (Actual)

PRIMARY OUTCOMES:
Logical reasoning test | 15 & 30 min inhalation and 5, 30, & 60 min post inhalation
Free recall memory test | 15 & 30 min inhalation and 5, 30, & 60 min post inhalation
Auditory reaction time | 15 & 30 min inhalation and 5,30 & 60 min post inhalation
Digit symbol substitution test | 2,15 & 30 min inhalation and 5,30 & 60 min post inhalation

CONTACTS AND LOCATIONS:
Overall Officials: James Zacny, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Anesthesia & Critical Care, Chicago, Illinois, United States

REFERENCES:
- [Background] Zacny JP, Yajnik S, Lichtor JL, Klafta JM, Young CJ, Thapar P, Rupani G, Coalson DW, Apfelbaum JL. The acute and residual effects of subanesthetic concentrations of isoflurane/nitrous oxide combinations on cognitive and psychomotor performance in healthy volunteers. Anesth Analg. 1996 Jan;82(1):153-7. doi: 10.1097/00000539-199601000-00028. PMID 8712393
- [Derived] Whelan J, Hackshaw A, McTiernan A, Grimer R, Spooner D, Bate J, Ranft A, Paulussen M, Juergens H, Craft A, Lewis I. Survival is influenced by approaches to local treatment of Ewing sarcoma within an international randomised controlled trial: analysis of EICESS-92. Clin Sarcoma Res. 2018 Mar 30;8:6. doi: 10.1186/s13569-018-0093-y. eCollection 2018. PMID 29610659